CLINICAL TRIAL: NCT03118999
Title: Plasma Level of Various Omega-3 Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 16.18.BIO
Record Dates: First submitted 2017-03-30; First posted 2017-04-18 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Single center, open design, randomized, controlled, cross-over trial with 3 test periods and 3 food supplements containing omega3 (one test period per product).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OM3-FFA (Experimental): Omega3 linked to free fatty acids
  Interventions: Dietary Supplement: OM3-MAG; Dietary Supplement: OM3-EE
- OM3 -MAG (Experimental): Omega3 linked to Monoacylglycerol
  Interventions: Dietary Supplement: OM3-FFA; Dietary Supplement: OM3-EE
- OM3-EE (Experimental): Omega3 linked to ethylester
  Interventions: Dietary Supplement: OM3-FFA; Dietary Supplement: OM3-MAG

INTERVENTIONS:
Dietary Supplement: OM3-FFA — Comparison of the effects of OM3-FFA versus OM3-MAG and OM3-EE in a crossover design
  Arms: OM3 -MAG; OM3-EE
Dietary Supplement: OM3-MAG — Comparison of the effects of OM3-MAG versus OM3-FFA and OM3-EE in a crossover design
  Arms: OM3-EE; OM3-FFA
Dietary Supplement: OM3-EE — Comparison of the effects of OM3-EE versus OM3-FFA and OM3-MAG in a crossover design
  Arms: OM3 -MAG; OM3-FFA

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetic properties of 3 OM3 oils after a single-dose administration in healthy volunteers

DETAILED DESCRIPTION:
This is a single center, open design, randomized, controlled, cross-over trial with 3 test periods and 3 products (one test period per product). The three different test periods will be separated by a washout period of at least 6 days (up to 21 days).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years old
* BMI in the normal and overweight range (18.5 to 29.9 kg/m2)
* Able to understand and to sign written informed consent prior to trial entry
* Informed consent signed

Exclusion Criteria:

* Food allergy
* Documented clinically relevant disease impacting the endpoints of the study or the safety of the subject, as determined by the medical (screening) visit:

  i. Malabsorptive disorders including but not limited to pancreatitis, Crohn's disease, etc. ii. Known hypertriglyceridemia (on anamnesis) iii. Known Type2 Diabetes Mellitus
* Under medication that may impact:

  1. Dietary fat absorption and metabolism like statins, bile acid sequestrants, lipid lowering medications, or fibrates (to the opinion of the investigator)
  2. Coagulation (blood thinning medications, anticoagulants). Indeed, OM3 have been shown to possibly exert some bleeding by themselves that may increase the bleeding effects of aspirin and anticoagulants
* Having taken omega-3, EPA/DHA, fish oil supplementation for more than two consecutive weeks during the last 2 months
* Having given blood within the last month, or willing to make a blood donation until one month following the end of the study
* Subjects not willing and/or not able to comply with scheduled visits and with the requirements of the study protocol, including trial products consumption and food restriction
* Pregnancy (on anamnesis)
* Any direct collaborator of the study leader (Dr. Maurice Beaumont)
* Currently participating or having participated in another clinical trial during the last month prior to the beginning of this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
AUC(0-24h) Plasma OM3 | From Time 0 hour to Time 24 hours
  Baseline-adjusted total plasma OM3 AUC(0-24h)

SECONDARY OUTCOMES:
Pharmacokinetic parameters (AUC) for EPA and DHA | From Time 0 hour to Time 24 hours
  AUC(0-24h) Plasma EPA and DHA
Pharmacokinetic parameters (Cmax) for EPA and DHA | From Time 0 hour to Time 24 hours
  Cmax Plasma EPA and DHA
Pharmacokinetic parameters (Tmax) for EPA and DHA | From Time 0 hour to Time 24 hours
  Tmax Plasma EPA and DHA

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Cuénoud, Study Director — Nestec Ltd.
Locations (1):
- Nestlé Research Center / Clinical Development Unit / Metabolic Unit, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No